CLINICAL TRIAL: NCT00507455
Title: A Phase 2, Randomized, Double-Blind, Parallel Group, Placebo Controlled, Multi-Center Study to Evaluate the Safety of the Co-administration of Solifenacin Succinate With 0.4 mg Tamsulosin Hydrochloride OCAS (TOCAS) Using Urodynamics in Male Subjects With Lower Urinary Tract Symptoms (LUTS) and Bladder Outlet Obstruction (BOO)
Brief Title: Solifenacin Succinate With Tamsulosin HCl in Males With Lower Urinary Tract Symptoms and Bladder Outlet Obstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 905-CL-058; 2007-001268-57 (EudraCT Number)
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Lower Urinary Tract Symptoms; Bladder Outlet Obstruction
Keywords: Lower Urinary Tract Symptoms; Bladder Outlet Obstruction; Treatment; Solifenacin Succinate; Tamsulosin hydrochloride
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder Neck Obstruction | interventions — Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received once daily, oral doses of placebo matching solifenacin succinate and tamsulosin tablets for 12 weeks.
  Interventions: Drug: Placebo to solifenacin; Drug: Placebo to tamsulosin
- 6 mg Solifenacin + 0.4 mg Tamsulosin (Experimental): Participants received once daily, oral doses of 6 mg solifenacin succinate and 0.4 mg tamsulosin tablets for 12 weeks.
  Interventions: Drug: solifenacin succinate; Drug: tamsulosin hydrochloride
- 9 mg Solifenacin + 0.4 mg Tamsulosin (Experimental): Participants received once daily, oral doses of 9 mg solifenacin succinate and 0.4 mg tamsulosin tablets for 12 weeks.
  Interventions: Drug: solifenacin succinate; Drug: tamsulosin hydrochloride

INTERVENTIONS:
Drug: solifenacin succinate — Solifenacin succinate tablets
  Other Names: YM905; VESIcare
  Arms: 6 mg Solifenacin + 0.4 mg Tamsulosin; 9 mg Solifenacin + 0.4 mg Tamsulosin
Drug: tamsulosin hydrochloride — Tamsulosin hydrochloride Oral Control Absorption System (TOCAS) tablets
  Other Names: Omnic Ocas; Flomax CR
  Arms: 6 mg Solifenacin + 0.4 mg Tamsulosin; 9 mg Solifenacin + 0.4 mg Tamsulosin
Drug: Placebo to solifenacin
  Arms: Placebo
Drug: Placebo to tamsulosin
  Arms: Placebo

SUMMARY:
A study to evaluate the safety of the co-administration of solifenacin succinate with tamsulosin hydrochloride in men with lower urinary tract symptoms (LUTS) and bladder outlet obstruction (BOO).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Lower Urinary Tract Symptoms (LUTS) and Bladder Outlet Obstruction (BOO)
* BOO indication by a Bladder Outlet Obstruction Index (BOOI) ≥ 20
* Patient has a total International Prostate Symptom Score (IPPS) score of ≥ 8 (Inclusion criteria for Baseline also)
* Patient had a maximum urinary flow rate of ≤ 12 mL/sec, with a voided volume of ≥ 120 mL during free flow in a representative assessment of uroflowmetry.

Exclusion Criteria:

* History of urinary retention in preceding 12 months
* Current urinary tract infection (UTI) or symptomatic and recurrent UTI of > 3 episodes within 12 months.
* Known clinical history or diagnosis of chronic inflammation, stone in bladder or ureter, or other causes of outflow tract obstruction
* Known diagnosis or history of carcinoma or previous pelvic radiation therapy, except non-metastatic basal or squamous cell carcinoma of the skin that had been treated successfully
* Clinically significant cardiovascular or cerebrovascular diseases within 6 months prior to Visit 1

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (33):
- United States (17):
  - Homewood, Alabama
  - La Mesa, California
  - Long Beach, California
  - San Bernardino, California
  - San Diego, California
  - Middlebury, Connecticut
  - New Port Richey, Florida
  - Coeur d'Alene, Idaho
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Watertown, Massachusetts
  - Las Vegas, Nevada
  - New York, New York
  - Greensboro, North Carolina
  - Austin, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
- Belgium (2):
  - Edegem
  - Kortrijk
- Czechia (3):
  - Olomouc
  - Pilsen
  - Prague
- Germany (4):
  - Aachen
  - Hagenow
  - Landshut
  - Mülheim
- Hungary (3):
  - Budapest
  - Szeged
  - Szekszárd
- Poland (4):
  - Bialystok
  - Mysłowice
  - Szczecin
  - Warsaw

REFERENCES:
- [Result] Kaplan SA, He W, Koltun WD, Cummings J, Schneider T, Fakhoury A. Solifenacin plus tamsulosin combination treatment in men with lower urinary tract symptoms and bladder outlet obstruction: a randomized controlled trial. Eur Urol. 2013 Jan;63(1):158-65. doi: 10.1016/j.eururo.2012.07.003. Epub 2012 Jul 17. PMID 22831853

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 mg Solifenacin + 0.4 mg Tamsulosin: Participants received once daily oral doses of 6 mg solifenacin succinate and 0.4 mg tamsulosin hydrochloride Oral Control Absorption System (TOCAS) tablets for 12 weeks.
- 9 mg Solifenacin + 0.4 mg Tamsulosin: Participants received once daily, oral doses of 9 mg solifenacin succinate and 0.4 mg tamsulosin hydrochloride Oral Control Absorption System (TOCAS)tablets for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Started | 74 | 74 | 74
Completed | 62 | 68 | 62
Not Completed | 12 | 6 | 12
Not completed — Adverse Event | 3 | 3 | 6
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Protocol Violation | 4 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Other - miscellaneous reason | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin | Total
Number analyzed (Participants) | 74 | 74 | 74 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (7.60) | 63.8 (8.43) | 65.6 (8.26) | 64.6 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 74 | 74 | 74 | 222
Race/Ethnicity, Customized [Number; unit: participants]
  White | 71 | 74 | 69 | 214
  Black or African-American | 2 | 0 | 2 | 4
  Asian | 1 | 0 | 1 | 2
  Other | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Non Hispanic or Latino | 72 | 71 | 69 | 212
  Hispanic or Latino | 2 | 3 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment in Detrusor Pressure at Maximum Flow Rate (PdetQmax)
Description: Detrusor pressure (Pdet) measures the force the detrusor muscle is exerting. This pressure is required to expel urine from the bladder during normal voiding. A high detrusor pressure may be observed in the presence of outflow tract obstruction. Detrusor pressure at maximum urinary flow rate (PdetQmax) was evaluated using simultaneous recording of urinary voiding by an uroflowmeter during detrusor pressure evaluation by cystometry.
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS) population consisted of participants who received at least one dose of double-blind treatment and had both urodynamic measurements at baseline and one or both measured at any post-baseline on-treatment visit. Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: cmH2O
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 60 | 67 | 58
cmH2O | -1.69 (3.15) | -7.84 (2.95) | -6.69 (3.20)
Statistical Analysis 1: Comparison: Placebo vs 6 mg Solifenacin + 0.4 mg Tamsulosin; A hierarchical step-down procedure was used to control for multiplicity. The comparison between solifenacin 6 mg + tamsulosin 0.4 mg and placebo was conducted first. If non-inferiority was demonstrated, solifenacin 9 mg + tamsulosin 0.4 mg was then compared to placebo. If the first comparison did not demonstrate non-inferiority, no further testing was performed. This procedure maintained the overall type I error of 1-sided 2.5%; Test type: Non-Inferiority or Equivalence — If the upper limit of the 2-sided 95% confidence interval (CI) for the difference from placebo was less than 15 cmH2O for PdetQmax, then the treatment is non-inferior to the placebo in PdetQmax; LS Mean Difference = -6.15, 95% CI 2-sided [-14.67 to 2.37] — Least squares (LS) means were analyzed using analysis of covariance (ANCOVA) with the site and treatment group as the factors and the baseline value as the covariate
Statistical Analysis 2: Comparison: Placebo vs 9 mg Solifenacin + 0.4 mg Tamsulosin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS Mean Difference = -5.00, 95% CI 2-sided [-13.85 to 3.84] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Post Void Residual Volume (PVR)
Description: Healthy micturitions result in complete emptying of the bladder. Post Void Residual (PVR) is the volume of urine retained after voiding (post-void residual urine). Post void residual volume was assessed by abdominal ultrasound. An increasing PVR over time is an indicator of abnormal bladder function or detrusor decompensation.
  End-of-treatment is the last post-baseline assessment during the treatment period.
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set (FAS) population with available data at each time point (as indicated by "N"). End of treatment includes participants who did not complete the Week 12 visit using the last observation carried forward method.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
mL
  Week 2 (N=61, 67, 58) | -10.21 (6.912) | 16.78 (6.525) | 8.97 (7.015)
  Week 4 (N=60, 67, 59) | -7.86 (6.225) | 14.92 (5.830) | 9.65 (6.229)
  Week 8 (N=58, 66, 58) | -12.44 (6.434) | 9.64 (5.950) | 6.64 (6.373)
  Week 12 (N=57, 63, 57) | 1.16 (7.346) | 26.81 (6.843) | 18.72 (7.244)
  End of Treatment (N=62, 67, 59) | 0.14 (6.809) | 25.63 (6.477) | 19.07 (6.923)

3. Primary Outcome: Change From Baseline to End of Treatment in Maximum Flow Rate (Qmax)
Description: The maximum flow rate (Qmax) during a micturition (urination) was recorded using uroflowmetry. A reduction in maximum flow rate may be due to an obstruction of the bladder outlet or a failure of the detrusor muscle to aid in expelling urine.
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS) population consisted of participants who received at least one dose of double-blind treatment and had urodynamic measurements at baseline and post-baseline on-treatment visit. Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: mL/sec
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
mL/sec | 0.17 (0.43) | 1.85 (0.41) | 2.35 (0.43)
Statistical Analysis 1: Comparison: Placebo vs 6 mg Solifenacin + 0.4 mg Tamsulosin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — If the lower limit of the 2-sided 95% confidence interval (CI) for the difference from placebo was greater than -3 mL/sec for Qmax, then the treatment is non-inferior to the placebo in Qmax; LS Mean Difference = 1.67, 95% CI 2-sided [0.50 to 2.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 9 mg Solifenacin + 0.4 mg Tamsulosin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; LS Mean Difference = 2.18, 95% CI 2-sided [0.98 to 3.37] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline to End of Treatment in Bladder Contractility Index (BCI)
Description: The Bladder Contractility Index (BCI) is a value used to measure the degree of contractility. BCI was calculated using the following formula:
  BCI = pdetQmax + 5Qmax.
  Strong contractility is a BCI > 150, normal contractility is a BCI of 100-150 and weak contractility is a BCI of < 100.
  LS means were adjusted for pooled center and Baseline value.
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS) population; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 60 | 67 | 58
units on a scale | -1.63 (3.705) | 1.84 (3.475) | 3.86 (3.764)

5. Secondary Outcome: Change From Baseline to End of Treatment in Percent Bladder Voiding Efficiency (BVE)
Description: Percent Bladder Voiding Efficiency (BVE) is a product of bladder contractility against the urethral resistance and is measured according to the degree of bladder emptying. BVE is expressed as a percentage and is calculated using the formula:
  Bladder Voiding efficiency = (Voided volume x 100)/maximum cystometric capacity.
  A higher number indicates a higher voiding efficiency.
  LS means were adjusted for pooled center and Baseline value.
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS) population; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: Percent voiding efficiency
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
Percent voiding efficiency | -0.67 (2.757) | -1.38 (2.634) | -3.79 (2.812)

6. Secondary Outcome: Safety Assessed by Adverse Events (AEs), Electrocardiogram (ECG), Vital Signs, Physical Exam and Laboratory Tests
Description: Abnormal laboratory parameters, vital signs or ECG data were defined as AEs if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A serious AE was an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important. AEs were assessed by the Investigator for intensity as mild (no disruption of normal daily activities), moderate (affected normal daily activities) or severe (inability to perform daily activities) and for causal relationship to study drug.
Time Frame: From first dose to within 30 days after last dose of double blind study medication (up to 16 weeks).
Population: Safety analysis set population consisted of participants who received at least 1 dose of double-blind treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 74 | 74 | 74
participants
  Any adverse event | 29 | 38 | 37
  Mild adverse event | 21 | 21 | 20
  Moderate adverse event | 6 | 13 | 12
  Severe adverse event | 2 | 4 | 5
  Serious adverse event | 1 | 2 | 2
  AE leading to study drug discontinuation | 3 | 3 | 6
  Drug-related adverse events | 15 | 24 | 26
  Deaths | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in International Prostate Symptoms Score (IPSS)
Description: The IPSS is a validated global questionnaire used to assess the degree of "bother" from benign prostatic hyperplasia symptoms and is based on the answers to 7 questions concerning urinary symptoms:
  * Sensation of incomplete emptying
  * Repeat urinating after 2 hours (frequency)
  * Start and stop several times (intermittency)
  * Urgency
  * Weak stream
  * Straining
  * Nocturia
  Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set (FAS) population with available data at each time point. End of treatment includes participants who did not complete the Week 12 visit using the last observation carried forward method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
units on a scale
  Week 2 (N=61, 67, 58) | -3.8 (0.58) | -4.5 (0.54) | -4.7 (0.59)
  Week 4 (N=60, 65, 57) | -5.3 (0.63) | -6.4 (0.59) | -6.2 (0.64)
  Week 8 (N=58, 67, 57) | -6.8 (0.74) | -7.1 (0.68) | -6.9 (0.74)
  Week 12 (N=58, 63, 57) | -6.9 (0.66) | -7.9 (0.62) | -7.2 (0.66)
  End of Treatment (N=62, 67, 59) | -6.6 (0.65) | -8.0 (0.62) | -6.9 (0.66)

8. Secondary Outcome: Change From Baseline in IPSS Voiding Score
Description: The IPSS is a validated global questionnaire used to assess the degree of "bother" from benign prostatic hyperplasia symptoms based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The voiding score is the sum of the responses to 4 questions relating to urination (incomplete emptying, intermittency, weak stream and straining) and ranges from 0 to 20 (asymptomatic to very symptomatic).
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
units on a scale
  Week 2 (N=61, 67, 58) | -2.2 (0.39) | -2.9 (0.37) | -2.6 (0.40)
  Week 4 (N=60, 65, 57) | -3.2 (0.45) | -3.8 (0.42) | -3.6 (0.46)
  Week 8 (N=58, 67, 57) | -4.1 (0.49) | -4.3 (0.45) | -3.8 (0.49)
  Week 12 (N=58, 64, 57) | -4.0 (0.45) | -4.7 (0.42) | -4.1 (0.45)
  End of Treatment (N=62, 67, 59) | -3.9 (0.44) | -4.6 (0.42) | -3.9 (0.45)

9. Secondary Outcome: Change From Baseline in IPSS Storage Score
Description: The IPSS is a validated global questionnaire used to assess the degree of "bother" from benign prostatic hyperplasia symptoms based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The storage symptom score is the sum of the responses to 3 questions relating to storage symptoms (frequency, urgency and nocturia) and ranges from 0 to 15 (asymptomatic to very symptomatic).
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
units on a scale
  Week 2 (N=62, 67, 58) | -1.5 (0.29) | -1.6 (0.27) | -2.1 (0.29)
  Week 4 (N=60, 66, 58) | -2.1 (0.30) | -2.6 (0.28) | -2.5 (0.30)
  Week 8 (N=58, 67, 58) | -2.7 (0.34) | -2.8 (0.31) | -3.1 (0.33)
  Week 12 (N=58, 63, 57) | -2.8 (0.30) | -3.3 (0.29) | -3.1 (0.30)
  End of Treatment (N=62, 67, 59) | -2.7 (0.30) | -3.4 (0.28) | -3.0 (0.30)

10. Secondary Outcome: Change From Baseline in Patient Perception of Bladder Condition (PPBC)
Description: The patient perception of bladder condition (PPBC) questionnaire asks participants to assess their bladder condition using a 6-point validated Likert scale which ranges from 1 (does not cause me any problems at all) to 6 (causes me many severe problems).
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
units on a scale
  Week 2 (N=61, 66, 58) | -0.5 (0.12) | -0.3 (0.11) | -0.5 (0.12)
  Week 4 (N=60, 66, 58) | -0.7 (0.13) | -0.5 (0.12) | -0.9 (0.13)
  Week 8 (N=58, 67, 58) | -1.0 (0.14) | -0.8 (0.13) | -1.1 (0.14)
  Week 12 (N=58, 64, 57) | -1.1 (0.14) | -1.0 (0.13) | -1.1 (0.14)
  End of Treatment (N=62, 67, 59) | -1.1 (0.13) | -0.9 (0.13) | -1.1 (0.14)

11. Secondary Outcome: Change From Baseline in Number of Micturitions Per 24 Hours
Description: A micturition is any voluntary urination, excluding episodes of incontinence only. The mean number of micturitions per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
micturitions
  Week 2 (N=60, 67, 59) | -0.44 (0.261) | -1.25 (0.243) | -1.19 (0.261)
  Week 4 (N=60, 65, 58) | -1.03 (0.285) | -1.32 (0.270) | -1.72 (0.287)
  Week 8 (N=58, 67, 58) | -1.33 (0.330) | -1.31 (0.302) | -2.00 (0.327)
  Week 12 (N=58, 65, 58) | -1.07 (0.333) | -1.91 (0.309) | -1.89 (0.330)
  End of Treatment (N=60, 67, 59) | -0.95 (0.328) | -1.91 (0.306) | -1.87 (0.328)

12. Secondary Outcome: Change From Baseline in Number of Urgency Episodes Per 24 Hours
Description: For each micturition and/or incontinence episode participants rated the degree of associated urgency (the sudden compelling desire to pass urine, which is difficult to defer) according to the following scale: 0: No Urgency, felt no need to empty my bladder but did so for another reason; 1: Mild urgency, could postpone passing water for as long as necessary; 2: Moderate urgency, could postpone passing water for a short while; 3: Severe urgency, could not postpone passing water; 4: Urge incontinence, leaked before reaching the toilet. An urgency episode is defined as an episode with urgency severity of three or higher.
  The mean number of urgency episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
urgency episodes
  Week 2 (N=60, 67, 59) | -0.59 (0.246) | -0.89 (0.230) | -0.95 (0.246)
  Week 4 (N=60, 65, 58) | -1.18 (0.254) | -1.39 (0.240) | -1.34 (0.255)
  Week 8 (N=58, 67, 58) | -1.45 (0.263) | -1.34 (0.241) | -1.08 (0.261)
  Week 12 (N=58, 65, 58) | -1.47 (0.247) | -1.54 (0.230) | -1.18 (0.245)
  End of Treatment (N=60, 67, 59) | -1.41 (0.249) | -1.45 (0.232) | -1.23 (0.249)

13. Secondary Outcome: Change From Baseline in Number of Incontinence Episodes Per 24 Hours
Description: The mean number of incontinence episodes (the involuntary leakage of urine) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Full analysis set (FAS) population who had 3-day averaged incontinence episodes >0 at Baseline and with available data at each time point. End of treatment includes participants who did not complete the Week 12 visit using the last observation carried forward method.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 13 | 10 | 13
incontinence episodes
  Week 2 (N=13, 10, 13) | -0.81 (0.368) | -1.45 (0.412) | -1.01 (0.352)
  Week 4 (N=13, 10, 13) | -1.00 (0.533) | -1.45 (0.596) | -0.81 (0.508)
  Week 8 (N=12, 10, 12) | -1.86 (0.489) | -1.55 (0.508) | -0.78 (0.453)
  Week 12 (N=12, 9, 12) | -1.99 (0.600) | -1.48 (0.654) | -0.85 (0.551)
  End of Treatment (N=13, 10, 13) | -1.54 (0.571) | -1.66 (0.639) | -1.02 (0.545)

14. Secondary Outcome: Change From Baseline in Volume Voided Per Micturition
Description: The mean volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 62 | 67 | 59
mL
  Week 2 (N=60, 67, 59) | 9.36 (4.415) | 31.46 (4.109) | 18.25 (4.408)
  Week 4 (N=60, 65, 58) | 10.40 (5.207) | 35.27 (4.920) | 30.34 (5.236)
  Week 8 (N=58, 67, 58) | 10.50 (6.125) | 33.72 (5.596) | 35.53 (6.064)
  Week 12 (N=58, 65, 58) | 9.03 (5.703) | 35.02 (5.283) | 31.18 (5.643)
  End of Treatment (N=60, 67, 59) | 7.56 (5.700) | 36.26 (5.305) | 30.33 (5.691)

15. Secondary Outcome: Change From Baseline in International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptom (ICIQ MLUTS) Total Symptom Score
Description: Male lower urinary tract symptoms were assessed by the ICIQ MLUTS questionnaire which consists of 13 questions regarding urinary symptoms. Each question is answered by the participant on a scale from 0 (never) to 4 (all the time). The total symptom score ranges from 0 to 52, where larger scores correspond to worse conditions.
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: Full analysis set (FAS) population with available data at Baseline and at each time point (indicated as "N"). End of treatment includes participants who did not complete the Week 12 visit using the last observation carried forward method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 60 | 66 | 57
units on a scale
  Week 4 (N=58, 66, 52) | -3.9 (0.60) | -4.5 (0.56) | -4.6 (0.64)
  Week 8 (N=55, 63, 53) | -5.5 (0.68) | -5.6 (0.63) | -5.8 (0.70)
  Week 12 (N=55, 61, 53) | -5.5 (0.70) | -6.5 (0.66) | -5.9 (0.71)
  End of Treatment (N=60, 66, 57) | -5.2 (0.69) | -6.0 (0.65) | -5.8 (0.71)

16. Secondary Outcome: Change From Baseline in ICIQ-MLUTS Total Symptom Bother Score
Description: The degree to which urinary symptoms bothered participants was assessed by the ICIQ MLUTS questionnaire which consists of 13 symptom bother questions. Each question is answered by the participant on a scale from 0 (not at all) to 10 (a great deal). The total bother score ranges from 0 to 130, where larger scores correspond to worse outcomes.
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 58 | 61 | 54
units on a scale
  Week 4 (N=52, 57, 48) | -14.6 (2.76) | -11.0 (2.62) | -17.0 (2.88)
  Week 8 (N=51, 55, 47) | -20.7 (2.88) | -19.4 (2.75) | -20.7 (3.01)
  Week 12 (N=51, 51, 47) | -22.6 (2.78) | -23.9 (2.74) | -23.9 (2.91)
  End of Treatment (N=58, 60, 53) | -21.7 (2.71) | -21.1 (2.65) | -22.4 (2.84)

17. Secondary Outcome: Change From Baseline in International Consultation on Incontinence Questionnaire - Lower Urinary Tract Symptom Quality of Life (ICIQ-LUTSqol) Symptom Score
Description: Quality of life was assessed by the ICIQ-LUTSqol questionnaire which consists of 19 questions regarding daily activities affected by urinary problems. Participants responded to each question on a scale from 1 (not at all) to 4 (a lot). The total symptom score ranges from 19 to 76, where larger scores correspond to a lesser quality of life).
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 40 | 44 | 39
units on a scale
  Week 4 (N=33, 36, 36) | -2.7 (0.93) | -2.4 (0.88) | -5.1 (0.88)
  Week 8 (N=33, 32, 31) | -3.6 (0.98) | -4.3 (0.99) | -6.7 (1.01)
  Week 12 (N=35, 33, 28) | -4.8 (1.10) | -6.5 (1.12) | -8.4 (1.21)
  End of Treatment (N=39, 39, 38) | -4.7 (1.05) | -5.3 (1.04) | -7.3 (1.05)

18. Secondary Outcome: Change From Baseline in ICIQ-LUTSqol Overall Symptom Interference of Life Score
Description: Participants were asked to rate how much their urinary symptoms interfered overall with their everyday life on a scale from 0 (not at all) to 10 (a great deal).
  Least squares (LS) means were adjusted for pooled center and the Baseline value.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Number analyzed (Participants) | 60 | 66 | 57
units on a scale
  Week 4 (N=57, 66, 56) | -1.2 (0.29) | -1.2 (0.27) | -1.3 (0.29)
  Week 8 (N=56, 65, 55) | -1.7 (0.29) | -1.7 (0.26) | -1.8 (0.29)
  Week 12 (N=56, 63, 55) | -2.1 (0.28) | -2.0 (0.26) | -2.2 (0.28)
  End of Treatment (N=60, 66, 57) | -2.0 (0.28) | -1.9 (0.26) | -2.1 (0.29)

ADVERSE EVENTS:
Time Frame: From first dose to within 30 days after last dose of double blind study medication (up to 16 weeks).
Arm/Group | Placebo | 6 mg Solifenacin + 0.4 mg Tamsulosin | 9 mg Solifenacin + 0.4 mg Tamsulosin
Serious Adverse Events (participants affected / at risk) | 1/74 | 2/74 | 2/74
Other Adverse Events (participants affected / at risk) | 10/74 | 17/74 | 19/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | 6 mg Solifenacin + 0.4 mg Tamsulosin (N=74) | 9 mg Solifenacin + 0.4 mg Tamsulosin (N=74)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Urethritis (Infections and infestations) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | 6 mg Solifenacin + 0.4 mg Tamsulosin (N=74) | 9 mg Solifenacin + 0.4 mg Tamsulosin (N=74)
Vision blurred (Eye disorders) | 1 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 3 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 9 | 14
Fatigue (General disorders) | 2 | 4 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 4
Headache (Nervous system disorders) | 6 | 3 | 2

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site only after Sponsor's prior written consent.